Official Title: Development and Preliminary Examination of Two Brief Personalized Feedback Interventions

Focused on Lab-based and EMA Alcohol Cues to Reduce Hazardous Young Adult Alcohol Use

Brief Title: Testing Brief Personalized Feedback Integrating EMA Alcohol Cue Information (Project ACE)

NCT number: NCT05373706

Document date: April 30, 2024

## STUDY PROTOCOL

Given the role of cue reactivity in eliciting alcohol-related cravings that can lead to increased alcohol use, the current study develops and tests a novel intervention strategy that may ultimately increase the strength of Personalized Feedback Intervention (PFI) effects to reduce young adult (YA) alcohol misuse. We developed a novel Cue Reactivity PFI based on Ecological Momentary Assessment (EMA) that will provide young adults with personalized feedback regarding the extent to which their urges to drink vary in response to alcohol cues. In turn, we anticipate that this feedback will increase young adults' awareness of this phenomenon and of personally relevant cues. The novel intervention provides strategies for handling craving in response to alcohol cues with the goal of reducing alcohol use resulting from alcohol-related cues.

The study design is a randomized clinical trial that includes online Ecological Momentary Assessments (EMAs) and online baseline, 2-week, and 3-month assessments. Participants are randomized to either a PFI condition or an assessment-only condition. The study tests initial development of the PFI intervention, which is in the form of personalized feedback regarding alcohol craving and is delivered online to the intervention group. All participants complete the EMA protocol (daily surveys 4x/day for 17 days), baseline, and 2-week and 3-month surveys. The online intervention is sent on Day 17 of the EMA protocol; therefore, the follow-ups are timed to occur 2-weeks and 3-months from Day 17.

Individuals who agreed to participate in the screening survey (Information Statement presented) and who were eligible based on the screening survey were contacted by research staff to verify their identity (e.g., name, date of birth). Participants were then sent a link to complete the informed consent process (Consent Form) and baseline survey. After participants completed the baseline survey, they were scheduled for an online, Zoom training session with a research staff member. In the Zoom session, participants first confirmed their identity by showing either a drivers license or ID card. Next, participants were shown a PowerPoint to aid in a discussion of the EMA survey process and study procedures. Upon completion of the Zoom training session, participants were randomized to either a cue reactivity PFI condition or assessment only condition.

All participants began their 17-day burst of EMA surveys on the first Friday after their Zoom session. Participants were sent one morning survey (between 7am and 12pm), and participants could choose the start of their 3-hour time block (e.g., 7-10am, 8-11am, or 9am-12pm). Participants were sent 3 afternoon/evening surveys (one survey in each three 2-hour time block: 1-3pm; 4-6pm; 7-9pm); afternoon/evening surveys were sent at the same time for every participant. Upon completion of this 17-day EMA period, participants in the intervention condition received access to their online personalized feedback and a brief survey to assess reactions to their feedback. The intervention material consists only of this one-time personalized feedback (accessible online) that is provided to participants after the 17-day EMA period. The feedback remains accessible after the first viewing if the participant chooses to view it again. All participants received a 2-week follow-up survey and a 3-month follow-up survey timed to occur 2 weeks and 3-months, respectively, from Day 17 of the EMA period.

Participants in the intervention condition can access their personalized feedback via an online link sent directly to them. The personalized feedback consists of pre-programmed content viewable on either a computer or mobile phone. The feedback content provides educational information about awareness of alcohol cues and how that awareness relates to alcohol use as well as summaries of the participants' own daily data that they completed during the EMA period.